CLINICAL TRIAL: NCT01685905
Title: Evaluation of the Usefulness of Interferon-γ Release Assays and Tuberculin Skin Test for Detection of Latent Mycobacterium Tuberculosis Infection in Korean Patients With Rheumatic Diseases
Brief Title: The Usefulness of Interferon-γ Release Assays and Tuberculin Skin Test for Detection of Latent Tuberculosis Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hanyang University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Sang-Cheol Bae, Professor, MD, PhD, MPH, Hanyang University
Other Study IDs: TST_IGRA
Record Dates: First submitted 2012-09-12; First posted 2012-09-14 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Rheumatic Disease; Rheumatoid Arthritis; Ankylosing Spondylitis; Tuberculosis
Keywords: rheumatic disease, latent tuberculosis
MeSH Terms: conditions — Rheumatic Diseases; Arthritis, Rheumatoid; Spondylitis, Ankylosing; Tuberculosis; Latent Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purposes of this study

1. to compare the positivity of tuberculin skin test(TST) and QuantiFERON-TB Gold (QFT-G), and determine the level of agreement between two tests in patients with rheumatic diseases
2. to evaluate the difference in the occurrence of active TB in patients who receive both QFT-G and TST compared with those who receive only TST for detecting of Latent tuberculosis infection(LTBI) who are candidates of TNF inhibitors.

DETAILED DESCRIPTION:
Study Assessment

1. The positive rates of QFT-G and TST as a screening test for LTBI

   * The positive rates of QFT-G and TST will be analyzed
   * Additional analysis will be performed according to the type of disease
2. The agreement between QFT-G and TST as a screening test for LTBI

   * The agreement between QFT-G and TST will be analyzed for patients with rheumatic diseases who examined both QFT-G and TST
   * Additional analysis will be performed according to the type of disease
3. The correlation of the occurrence of active TB and two tests (QFT-G and TST)

   * The analysis of the correlation of the occurrence of active TB and two tests will be conducted for patients who have experienced anti-TNF agents

3-1. The occurrence of active TB in accordance with results of TST

3-2. The occurrence of active TB in accordance with results of QFT-G

3-3. The difference in the occurrence of active TB in patients performed both QFT-G and TST compared with those performed only TST for detecting of LTBI who are candidates of TNF inhibitors (pilot study).

ELIGIBILITY:
Inclusion Criteria:

* patients with rheumatic diseases who examined TST or QFT-G in Hanyang university hospital from 2004 to 2010

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1) Estimation of the positive rates and agreement between QFT-G and TST
  * Approximately 2,000 patients with rheumatic diseases who examined TST or QFT-G in Hanyang university hospital from 2004 to 2010 2) Determining the difference in the occurrence of active TB in the TNF inhibitor user according to the screening and the treatment of LTBI.
  * Approximately 400 patients with rheumatic diseases who received TST or QFT-G before using anti-TNF agents in Hanyang university hospital from 2004 to 2010
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
The agreement between QuantiFERON-TB Gold(QFT-G) and tuberculin skin test(TST) as a screening test for latent tuberculosis infection(LTBI) | one year

SECONDARY OUTCOMES:
The correlation of the occurrence of active Tuberculosis and two tests (QuantiFERON-TB Gold (QFT-G) and tuberculosis skin test(TST)) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Sang-cheol Bae, director, Principal Investigator — Hanyang University Hospital for Rheumatic Disease
Locations (1):
- Hanyang University Hospital for rheumatic disease, Seoul, Sung-dong Gu, South Korea